CLINICAL TRIAL: NCT02389569
Title: A Prospective, Double-blind, Randomized, Group Controlled Clinical Study on the Use of Biosilicate Under Resin Composite Restorations in Caries Affected Teeth
Brief Title: Clinical Study of Biosilicate Under Resin Composite Restorations in Caries Affected Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Karen Pintado Palomino, MSc, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE nº: 27790214.1.0000.541
Record Dates: First submitted 2015-02-24; First posted 2015-03-17 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Dental Caries
Keywords: Biomaterial; Dental caries; Composite
MeSH Terms: conditions — Dental Caries | interventions — inzoma; Vivadent; sodium oxide-calcium oxide-silicon dioxide-diphosphorus pentoxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Adhesive system treatment (Experimental): Four groups ( Two will be treat with Etch-and-Rinse Adhesive System and two will be treated with two step Self-Etch Adhesive System).
  Interventions: Procedure: Adhesive system
- Restoration protocol (Experimental): Four groups ( Two will be treat with experimental Biosilicate and two will be the control groups).
  Interventions: Procedure: Restoration protocol

INTERVENTIONS:
Procedure: Adhesive system — Etch-and-rinse and Self-etch adhesive system will be applied in volunteers that received different types of restoration protocol.
  Other Names: Etch-and-rinse adhesive: Adper Single bond (3M, Brazil); Self-etch: Adhese (2 step self-etch) (Ivoclar, Vivadent)
  Arms: Adhesive system treatment
Procedure: Restoration protocol — Volunteers will be treated by two types of protocol restoration : 1) Biosilicate (powder) or 2) Control (without Biosilicate). In sequence, adhesive (self-etch or etch and rinse) and composite resin will be used for restoration.
  Other Names: Biosilicate (Vitrovita, Brazil); Control
  Arms: Restoration protocol

SUMMARY:
This study aimed to evaluate the clinical performance of a novel vitro-ceramic biomaterial (Biosilicate®) as treatment of caries-affected dentin in posterior resin restorations. A total of 94 restorations of 66 participants were selected and assigned at random into four groups: 1 (Biosilicate / Two-step etch and rinse system), 2 (Control / Two-step etch and rinse system), 3 (Biosilicate / Two-step self-etching system) and 4 (Control / Two-step self-etching system). Two operators carried out the adhesive protocols and restored the cavities with a nano-hybrid resin composite (IPS Empress, Ivoclar) using the incremental technique. Participants were recalled at one week, 6, 12 and 18 months for clinical evaluation performed by two blinders and calibrated examiners according FDI criteria.

DETAILED DESCRIPTION:
Background: Dental caries has decreased in recent years, but is still the main oral health problem in developed and undeveloped industrialized countries. The purpose of this study is to evaluate clinical performance of resin-based composite Class I and II restorations in association with Biosilicate.

Methods: Eighty patients with carious lesions will be receive restorations in premolars and molars, which will be randomly allocated in four experimental groups: G1 (Biosilicate, AdperSingle Bond 2 and IPS Empress Direct composite), G2 (Adper Single Bond 2 and IPS Empress Direct composite), G3 (Biosilicate, AdheSe and IPS Empress Direct composite) e G4 (AdheSE and IPS Empress Direct composite) To participate in the clinical trial, qualified subjects must meet for inclusion and exclusion criteria. Sixty-four (64) selected volunteers will be fully informed on the nature of the study and after had signed a Term of Acceptance defined by the Ethics Committee (FORP - USP), they will be invited to participate.

Carious teeth will be cleaned with a pumice-water slurry and rubber cup to remove salivary pellicle and any bacterial plaque. As much as possible, local anesthesia will be. After caries removal (high and low-speed handpieces under abundant water irrigation), patients will be allocated randomly in the four experimental groups cited above. Final contouring and polishing of the restorations will be performed at the same appointment, using a fine-grit diamond bur (KG Sorensen), silicon carbide polisher (Viking Kit, KG Sorensen), silicone rubber tips (Viking Kit, KG Sorensen) flexible discs (Sof-Lex, 3M ESPE), and polishing pastes (Diamond Excel, FGM).

Two trained and calibrated evaluators, fully blinded to the restorative techniques used, will be evaluating the restorations at baseline (one week after placement of restorations), after 06, 12 and 18 months using FDI criteria. All restorations will be photographed at every evaluation point. Esthetic, Functional and Biological proprieties will be used as key parameters determining the overall clinical success. Data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Cavitated or non-cavitated active carious lesions in dentin (Class I and/or II)
* Carious lesion in teeth with or without restoration in at least one tooth (upper or lower premolar and/or molar).
* No history of spontaneous pain
* Pulp vital tests positive
* No evidence of periapical radiolucency

Exclusion Criteria:

* Compromised medical history
* Periodontal disease
* Pulp necrosis
* Absence of antagonist teeth
* Severe bruxism
* Active orthodontic treatment
* Teeth with cracks and premature contact.
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Primary Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance of Biosilicate in caries lesion using FDI evaluation criteria | 18 months
  Two experienced and calibrated dentists, not involved with the placement of the restorations will be assess the efficiency of Biosilicate under composite restoration of Class I and Class II dentin caries lesions by record instrument to record the esthetic, functional and biological properties over a 18 months time frame. These variables will be ranked according to the FDI criteria in the following scores: clinically very good, clinically good, clinically sufficient/ satisfactory, clinically unsatisfactory and clinically poor.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Pintado Palomino, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirao Preto Campus, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Dental School of Ribeirão Preto website — http://www.forp.usp.br